CLINICAL TRIAL: NCT00035295
Title: A Double-Blind, Multicenter, Placebo-and Active-Controlled Acute and Extension Study of 2 Doses of MK-0869 in the Treatment of Patients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-061)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-061; 2006_404
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0869, aprepitant
Drug: Comparator: placebo

SUMMARY:
A clinical study to determine the efficacy and safety of an Treatment of MK0869

in the treatment of depression.

DETAILED DESCRIPTION:
The duration of treatment is 8 weeks.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2001-11-08 (Actual); Primary Completion 2003-12-05 (Actual); Study Completion 2003-12-05 (Actual)

PRIMARY OUTCOMES:
HAMD-17 total score at week 8. Tolerability.

SECONDARY OUTCOMES:
CGI-I score at week 8, at least 50% reduction in the HAMD-17 total score, and Sheehan Disability Score at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Keller M, Montgomery S, Ball W, Morrison M, Snavely D, Liu G, Hargreaves R, Hietala J, Lines C, Beebe K, Reines S. Lack of efficacy of the substance p (neurokinin1 receptor) antagonist aprepitant in the treatment of major depressive disorder. Biol Psychiatry. 2006 Feb 1;59(3):216-23. doi: 10.1016/j.biopsych.2005.07.013. Epub 2005 Oct 24. PMID 16248986
- [Background] Liu KS, Snavely DB, Ball WA, Lines CR, Reines SA, Potter WZ. Is bigger better for depression trials? J Psychiatr Res. 2008 Jul;42(8):622-30. doi: 10.1016/j.jpsychires.2007.07.003. Epub 2007 Sep 7. PMID 17825841
- Available data/document: CSR Snyopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html